CLINICAL TRIAL: NCT05556330
Title: Assessment of Horizontal Ridge Augmentation in Anterior Mandible Using Computer Guided Autogenous Cortical Shell Technique Versus Free Hand Technique: Randomized Clinical Trial
Brief Title: Computer Guided Versus Free Hand Horizontal Ridge Augmentation in Anterior Mandible.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Sakr, OMFS Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13522
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Computer Guided Alveolar Bone Augmentaion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- horizontal ridge augmentation by computer guided autogenous cortical shell technique (Experimental)
  Interventions: Procedure: computer guided autogenous cortical shell technique
- horizontal ridge augmentation by free hand autogenous cortical shell technique (Active Comparator)
  Interventions: Procedure: computer guided autogenous cortical shell technique

INTERVENTIONS:
Procedure: computer guided autogenous cortical shell technique — computer guided autogenous cortical shell technique

SUMMARY:
Assessment of horizontal ridge augmentation in anterior mandible using computer guided autogenous cortical shell technique versus free hand technique:

randomized clinical trial

DETAILED DESCRIPTION:
patients with deficient anterior mandible were included in this study where control group patients received free hand harvesting and fixation of cortical shells from the symphysis, while the study group patients received the same protocol using 2 patient specific guides (psg) the first guide used for safe and accurate graft harvesting with the proposed dimensions while the second guide used for shell fixation leaving the desired gap with the recipient site that was filled with a particulate mix of xeno and auto grafts .the first guide was fixed in place allowing for accurate harvesting of the cortical shell of desired dimensions from the symphysis Then; the harvested shell was fixed to the second guide outside the patients mouth using micro screws And this fixation guide was finally secured to its final position using two interlocking wings to lock into the first guide at the surgical site as a verification step for the accuracy of the whole procedure. Finally, the 2 guides were removed after shell fixation to the recipient site in a through and through manner st the proposed planed position.

ELIGIBILITY:
Inclusion Criteria:

* • Age ranges from 25-55 years. No sex predilection.

  * Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
  * Edentulous anterior mandible with horizontally deficient alveolar ridge that is less than 3mm width.
  * Normal vertical dimension with normal inter-arch space.
  * The minimum number of missing teeth in the anterior mandible alveolar ridge is two adjacent teeth.

Exclusion Criteria:

* • Intra-bony lesions (e.g., cysts) or infections (e.g., abscess) that may retard the osteotomy healing.

  * Previous grafting procedures in the edentulous area.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge horizontal bone gain | one day
  amount of horizontal bone gain in millimeters measured by cbct

SECONDARY OUTCOMES:
Alveolar ridge horizontal augmentation accuracy in 3D space | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No